CLINICAL TRIAL: NCT06816524
Title: The Effects of Iron Treatment on Malaria and Measles Vaccine Response in Kenyan Infants With Iron Deficiency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Stoffel (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other); University of Oxford - Nuffield Department of Orthopaedics, Rheumatology and Musculoskeletal Sciences (Unknown); Faculty of Medical Sciences, Radboud University of Medical Center (Unknown); National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Sponsor-Investigator, Nicole Stoffel, Prof., ETH Zurich
Organization: ETH Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MEMA
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Iron Deficiencies
Keywords: Iron deficiency; Vaccine immunogenicity; Malaria; Measles
MeSH Terms: conditions — Iron Deficiencies; Malaria; Measles | interventions — Malaria Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron treatment group (Active Comparator): daily multivitamin + daily iron syrup from age 6 to 10 months
  Interventions: Dietary Supplement: Iron syrup; Dietary Supplement: Multivitamin syrup; Biological: R21-Matrix/M Vaccine (malaria vaccine); Biological: Measles-Rubella vaccine
- Control group (Other): daily multivitamin syrup from age 6 to 10 months
  Interventions: Dietary Supplement: Multivitamin syrup; Biological: R21-Matrix/M Vaccine (malaria vaccine); Biological: Measles-Rubella vaccine

INTERVENTIONS:
Dietary Supplement: Iron syrup — Iron syrup administered daily from 6 to 10 months of age.
  Arms: Iron treatment group
Dietary Supplement: Multivitamin syrup — Multivitamin syrup administered daily from 6 to 10 months of age.
Biological: R21-Matrix/M Vaccine (malaria vaccine) — R21-Matrix/M vaccine administered in 3 doses at 7, 8 and 9 months of age.
Biological: Measles-Rubella vaccine — Measles-Rubella vaccine administered at 9 months of age.

SUMMARY:
Malaria and iron deficiency cause a significant burden of disease in Africa. Iron deficiency (ID) might affect immune responses to vaccination.

In this double-blind randomized controlled trial, we aim to assess: (1) whether ID impairs R21/Matrix-M and measles (MR) vaccine response, (2) whether iron treatment at time of vaccination improves vaccine response.

ELIGIBILITY:
Inclusion Criteria:

* Subject's caregiver is willing and able to give informed consent
* Male or Female, 6 months (+/- 2 weeks) of age
* Mother at least ≥15 years of age
* Iron deficient (erythrocyte zinc protoporphyrin (ZnPP) >61 μmol/mol heme)
* With or without anemia (anemia defined by Hb <110 g/L)

Exclusion Criteria:

* Severely anemic (Hb <70 g/L)
* Malaria vaccination prior to enrollment
* Medical condition that precludes study involvement
* Iron supplementation 2 weeks before enrollment
* Acute or chronic infection (e.g. HIV)
* Wasted (length for height z score of ≥-2) or underweight (weight for age z score ≥-2).

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
NANP-specific IgG | At 10 months of age (1 month after the 3rd R21/Matrix-M dose)
  NANP-specific IgG
anti- full lengths CSP IgG | At 10 months of age (1 month after the 3rd R21/Matrix-M dose)
  anti- full lenghts circumsporozoite protein IgG
anti- C-terminal CSP IgG | At 10 months of age (1 month after the 3rd R21/Matrix-M dose)
  anti- full lenghts circumsporozoite protein IgG
anti-measles IgG | At 10 months of age (1 month after the first MR dose)
  anti-measles IgG titre

SECONDARY OUTCOMES:
NANP-specific IgG | At 8 months age (1 month after the first R21/Matrix-M dose)
  NANP-specific IgG
NANP-specific IgG | At 9 months age (1 month after the second R21/Matrix-M dose)
  NANP-specific IgG
anti- full lengths CSP IgG | At 8 months age (1 month after the first R21/Matrix-M dose)
  anti- full lengths circumsporozoite protein IgG
anti- full lengths CSP IgG | At 9 months age (1 month after the second R21/Matrix-M dose)
  anti- full lengths circumsporozoite protein IgG
anti-CSP IgA | At 8 months age (1 month after the first R21/Matrix-M dose)
  anti- circumsporozoite protein IgA titre
anti-CSP IgA | At 9 months age (1 month after the second R21/Matrix-M dose)
  anti-circumsporozoite protein IgA titre
anti-CSP IgM | At 8 months age (1 month after the first R21/Matrix-M dose)
  anti circumsporozoite protein IgM titre
anti-CSP IgM | At 9 months age (1 month after the second R21/Matrix-M dose)
  anti-circumsporozoite protein IgM titre
Haemoglobin | 6 months of age
  Haemoglobin concentration (g/dL)
Haemoglobin | 7 months of age
  Haemoglobin concentration (g/dL)
Haemoglobin | 8 months of age
  Haemoglobin concentration (g/dL)
Haemoglobin | 9 months of age
  Haemoglobin concentration (g/dL)
Haemoglobin | 10 months of age
  Haemoglobin concentration (g/dL)
Plasma iron | 6 months of age
  Plasma iron concentration (μg/mL)
Plasma iron | 7 months of age
  Plasma iron concentration (μg/mL)
Plasma iron | 8 months of age
  Plasma iron concentration (μg/mL)
Plasma iron | 9 months of age
  Plasma iron concentration (μg/mL)
Plasma iron | 10 months of age
  Plasma iron concentration (μg/mL)
Total iron binding capacity | 6 months of age
  Total iron binding capacity (mcd/dL)
Total iron binding capacity | 7 months of age
  Total iron binding capacity (mcd/dL)
Total iron binding capacity | 8 months of age
  Total iron binding capacity (mcd/dL)
Total iron binding capacity | 9 months of age
  Total iron binding capacity (mcd/dL)
Total iron binding capacity | 10 months of age
  Total iron binding capacity (mcd/dL)
Transferrin saturation | 6 months of age
  Transferrin saturation (%)
Transferrin saturation | 7 months of age
  Transferrin saturation (%)
Transferrin saturation | 8 months of age
  Transferrin saturation (%)
Transferrin saturation | 9 months of age
  Transferrin saturation (%)
Transferrin saturation | 10 months of age
  Transferrin saturation (%)
Plasma Ferritin | 6 months of age
  Plasma Ferritin concentration (μg/mL)
Plasma Ferritin | 7 months of age
  Plasma Ferritin concentration (μg/mL)
Plasma Ferritin | 8 months of age
  Plasma Ferritin concentration (μg/mL)
Plasma Ferritin | 9 months of age
  Plasma Ferritin concentration (μg/mL)
Plasma Ferritin | 10 months of age
  Plasma Ferritin concentration (μg/mL)
Soluble transferrin receptor | 6 months of age
  Soluble transferrin receptor concentration (μg/mL)
Soluble transferrin receptor | 7 months of age
  Soluble transferrin receptor concentration (μg/mL)
Soluble transferrin receptor | 8 months of age
  Soluble transferrin receptor concentration (μg/mL)
Soluble transferrin receptor | 9 months of age
  Soluble transferrin receptor concentration (μg/mL)
Soluble transferrin receptor | 10 months of age
  Soluble transferrin receptor concentration (μg/mL)
C-reactive protein | 6 months of age
  C-reactive protein concentration (mg/L)
C-reactive protein | 7 months of age
  C-reactive protein concentration (mg/L)
C-reactive protein | 8 months of age
  C-reactive protein concentration (mg/L)
C-reactive protein | 9 months of age
  C-reactive protein concentration (mg/L)
C-reactive protein | 10 months of age
  C-reactive protein concentration (mg/L)
Retinol-binding protein | 6 months of age
  Retinol-binding protein concentration (μmol/L)
Retinol-binding protein | 7 months of age
  Retinol-binding protein concentration (μmol/L)
Retinol-binding protein | 8 months of age
  Retinol-binding protein concentration (μmol/L)
Retinol-binding protein | 9 months of age
  Retinol-binding protein concentration (μmol/L)
Retinol-binding protein | 10 months of age
  Retinol-binding protein concentration (μmol/L)
Alpha-glycoprotein | 6 months of age
  Alpha-glycoprotein concentration (g/L)
Alpha-glycoprotein | 7 months of age
  Alpha-glycoprotein concentration (g/L)
Alpha-glycoprotein | 8 months of age
  Alpha-glycoprotein concentration (g/L)
Alpha-glycoprotein | 9 months of age
  Alpha-glycoprotein concentration (g/L)
Alpha-glycoprotein | 10 months of age
  Alpha-glycoprotein concentration (g/L)
anti- C-terminal CSP IgG | At 8 months age (1 month after the first R21/Matrix-M dose)
  anti- C-terminal circumsporozoite protein IgG
anti- C-terminal CSP IgG | At 9 months age (1 month after the second R21/Matrix-M dose)
  anti- C-terminal circumsporozoite protein IgG
anti-CSP IgA | At 10 months age (1 month after the 3rd R21/Matrix-M dose)
  anti-circumsporozoite protein IgA titre
anti-CSP IgM | At 10 months age (1 month after the 3rd R21/Matrix-M dose)
  anti-circumsporozoite protein IgM titre
anti-measles IgG avidity | At 10 months age (1 month after the first MR dose)
  anti-measles IgG avidity

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stoffel, PhD, Principal Investigator — ETH Zurich

IPD SHARING:
Plan to Share IPD: No